CLINICAL TRIAL: NCT01088412
Title: The Genetics and Neuroendocrinology of Short Stature International Study (GeNeSIS)
Brief Title: Observational Study of Somatropin Treatment in Children
Acronym: GeNeSIS
Status: Completed | Type: Observational
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 2712; B9R-EW-GDFC (Other: ELI Lilly and Company)
Record Dates: First submitted 2010-02-25; First posted 2010-03-17 (Estimated); Results first posted 2019-05-13 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2018-07

CONDITIONS: Growth Hormone (GH) Deficiency; Short Stature Homeobox Containing Gene (SHOX) Deficiency; SHOX Deficiency-related Disorder; Non-GH-deficient Growth Disorders
MeSH Terms: interventions — Human Growth Hormone; DNA, Recombinant; DNA, Ribosomal; Growth Hormone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — If participant consented a DNA sample is kept until the end of the study
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Treated: Participants treated with somatropin for improvement of growth
  Interventions: Drug: Somatropin (recombinant deoxyribonucleic acid [rDNA] origin)
- Untreated: Untreated participants with presence or history of neoplastic disease evaluated for endocrine or growth disorder or with any SHOX deficiency related disorder

INTERVENTIONS:
Drug: Somatropin (recombinant deoxyribonucleic acid [rDNA] origin) — Dose, frequency and duration at discretion of attending physician.
  Other Names: Humatrope; LY137998
  Groups: Treated

SUMMARY:
GeNeSIS is an open-label, multinational, multicenter, observational study to evaluate the safety and effectiveness of Humatrope treatment.

GeNeSIS is a modular program that includes:

* Core study: Evaluating the safety and effectiveness of Humatrope in the observational setting
* Genetic Analysis Sub-study: Investigating the genetic defects underlying growth hormone (GH) deficiency and non-GH-deficient growth disorders
* Growth Prediction Sub-study: Working to validate and refine specific models to accurately predict growth response to GH
* Short Stature Homeobox containing gene (SHOX) Deficiency Sub-study: Elucidating the clinical, endocrine and radiological features of participants with SHOX deficiency due to loss of, or mutation in the SHOX gene (including participants with Turner syndrome)
* Neoplasia Sub-study: To characterize the natural history of neoplastic disease, especially in relation to recurrence/progression of primary neoplasia or development of secondary neoplasia in children with a history of neoplasia

ELIGIBILITY:
Inclusion Criteria:

All participants participating in GeNeSIS must be enrolled in the core study. Participants for whom written consent to release information is provided may enter the core study if they meet any of the following inclusion guidelines:

* Treatment with Humatrope for improvement of growth.
* No treatment with somatropin in participants with a history of neoplasia or in those with any SHOX deficiency-related disorder.

Exclusion Criteria:

* Participants with closed epiphyses are not eligible for GeNeSIS entry. However, participants may remain in the study if epiphyseal closure occurs during study participation.

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Clinics and private practices
Sampling Method: Non-Probability Sample
Enrollment: 22845 (Actual)
Dates: Start 1999-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company

REFERENCES:
- [Derived] Child CJ, Zimmermann AG, Chrousos GP, Cummings E, Deal CL, Hasegawa T, Jia N, Lawrence S, Linglart A, Loche S, Maghnie M, Perez Sanchez J, Polak M, Predieri B, Richter-Unruh A, Rosenfeld RG, Yeste D, Yorifuji T, Blum WF. Safety Outcomes During Pediatric GH Therapy: Final Results From the Prospective GeNeSIS Observational Program. J Clin Endocrinol Metab. 2019 Feb 1;104(2):379-389. doi: 10.1210/jc.2018-01189. PMID 30219920
- [Derived] Deal C, Kirsch S, Chanoine JP, Lawrence S, Cummings E, Rosolowsky ET, Marks SD, Jia N, Child CJ; GeNeSIS National Board on behalf of the GeNeSIS Canada Investigators. Growth hormone treatment of Canadian children: results from the GeNeSIS phase IV prospective observational study. CMAJ Open. 2018 Sep 10;6(3):E372-E383. doi: 10.9778/cmajo.20180020. Print 2018 Jul-Sep. PMID 30201821
- [Derived] Quigley CA, Child CJ, Zimmermann AG, Rosenfeld RG, Robison LL, Blum WF. Mortality in Children Receiving Growth Hormone Treatment of Growth Disorders: Data From the Genetics and Neuroendocrinology of Short Stature International Study. J Clin Endocrinol Metab. 2017 Sep 1;102(9):3195-3205. doi: 10.1210/jc.2017-00214. PMID 28575299
- [Derived] Blum WF, Deal C, Zimmermann AG, Shavrikova EP, Child CJ, Quigley CA, Drop SL, Cutler GB Jr, Rosenfeld RG. Development of additional pituitary hormone deficiencies in pediatric patients originally diagnosed with idiopathic isolated GH deficiency. Eur J Endocrinol. 2013 Nov 22;170(1):13-21. doi: 10.1530/EJE-13-0643. Print 2014 Jan. PMID 24088548
- [Derived] Deal C, Hasselmann C, Pfaffle RW, Zimmermann AG, Quigley CA, Child CJ, Shavrikova EP, Cutler GB Jr, Blum WF. Associations between pituitary imaging abnormalities and clinical and biochemical phenotypes in children with congenital growth hormone deficiency: data from an international observational study. Horm Res Paediatr. 2013;79(5):283-92. doi: 10.1159/000350829. Epub 2013 May 16. PMID 23689058
- [Derived] Child CJ, Zimmermann AG, Scott RS, Cutler GB Jr, Battelino T, Blum WF; GeNeSIS International Advisory Board. Prevalence and incidence of diabetes mellitus in GH-treated children and adolescents: analysis from the GeNeSIS observational research program. J Clin Endocrinol Metab. 2011 Jun;96(6):E1025-34. doi: 10.1210/jc.2010-3023. Epub 2011 Apr 13. PMID 21490076

RESULTS

PARTICIPANT FLOW:
Groups:
- Treated: Treatment with Humatrope for improvement of growth. Growth Hormone (GH) product.
- Untreated: No treatment with Humatrope in participants with a history of neoplasia or in those with any short stature homeobox containing gene (SHOX) deficiency-related disorder .
- FG002: Treatment with Humatrope unknown.
Period: Overall Study
Arm/Group | Treated | Untreated | FG002
Started | 22311 | 457 | 77
Safety Modified Evaluable (SME) | 22294 | 456 | 0
SME With at Least 1 Follow Up (FU) | 21178 | 306 | 0
SME+ >= 1 FU and Unknown Arm | 21177 | 306 | 40
SME+ >= 1 FU and No Previous Cancer | 20556 | 192 | 0
SME+ >= 1 FU and Previous Cancer | 622 | 114 | 0
Completed | 4294 | 21 | 5
Not Completed | 18017 | 436 | 72
Not completed — Adverse Event | 38 | 0 | 0
Not completed — Death | 42 | 6 | 0
Not completed — Other Reason per Case Report Form | 2089 | 103 | 9
Not completed — Withdrawal by Subject | 1761 | 25 | 1
Not completed — Received Another GH Product | 79 | 0 | 0
Not completed — Participant Moved | 601 | 21 | 2
Not completed — Physician Decision | 1041 | 8 | 4
Not completed — Sponsor Decision | 4467 | 79 | 23
Not completed — Third Party Required to Change Brand | 487 | 0 | 0
Not completed — Lost to Follow-up | 3052 | 130 | 11
Not completed — Study Summary Not Completed | 4360 | 64 | 22

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Treated: Treatment with Humatrope for improvement of growth.
- Untreated: No treatment with Humatrope in participants with a history of neoplasia or in those with any SHOX deficiency-related disorder.
- Unknown: Treatment with Humatrope unknown.
- Total: Total of all reporting groups
Arm/Group | Treated | Untreated | Unknown | Total
Number analyzed (Participants) | 22311 | 457 | 77 | 22845
Age, Customized [Number; unit: participants] — Age unavailable for 136 treated participants, 10 untreated participants, and 49 unknown participants.
  participants
    <=18 years | 21724 | 427 | 27 | 22178
    Between 18 and 65 years | 451 | 20 | 1 | 472
    >=65 years | 0 | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: participants] — No gender available for 32 treated participants, 1 untreated participant, and 49 unknown participants.
  participants
    Female | 8917 | 247 | 11 | 9175
    Male | 13362 | 209 | 17 | 13588
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 959 | 18 | 0 | 977
  Not Hispanic or Latino | 9279 | 166 | 0 | 9445
  Unknown or Not Reported | 12073 | 273 | 77 | 12423
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 0 | 0 | 9
  Asian | 260 | 3 | 0 | 263
  Native Hawaiian or Other Pacific Islander | 16 | 0 | 0 | 16
  Black or African American | 295 | 8 | 0 | 303
  White | 8328 | 148 | 0 | 8476
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 13403 | 298 | 77 | 13778
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 87 | 0 | 0 | 87
  Austria | 103 | 0 | 0 | 103
  Belgium | 83 | 0 | 0 | 83
  Canada | 850 | 17 | 3 | 870
  Czechia | 332 | 12 | 0 | 344
  Denmark | 5 | 0 | 1 | 6
  Finland | 28 | 0 | 0 | 28
  France | 1667 | 150 | 4 | 1821
  Germany | 2685 | 24 | 14 | 2723
  Greece | 290 | 14 | 1 | 305
  Hungary | 332 | 2 | 0 | 334
  Iceland | 48 | 0 | 0 | 48
  India | 212 | 30 | 0 | 242
  Italy | 771 | 13 | 4 | 788
  Japan | 2352 | 0 | 4 | 2356
  Kazakhstan | 29 | 0 | 0 | 29
  Lithuania | 90 | 0 | 0 | 90
  Netherlands | 317 | 0 | 3 | 320
  Norway | 8 | 0 | 0 | 8
  Pakistan | 172 | 6 | 0 | 178
  Russia | 180 | 15 | 0 | 195
  Singapore | 13 | 3 | 0 | 16
  Slovakia | 94 | 0 | 0 | 94
  South Africa | 106 | 1 | 2 | 109
  Spain | 1404 | 9 | 9 | 1422
  Sweden | 53 | 0 | 0 | 53
  Taiwan | 114 | 0 | 1 | 115
  Thailand | 33 | 0 | 0 | 33
  United Kingdom | 41 | 1 | 0 | 42
  United States | 9812 | 160 | 31 | 10003
Diagnostic Groups [Number; unit: participants]
  Chronic Renal Insufficiency (CRI) | 87 | 0 | 0 | 87
  Growth Hormone Deficiency (GHD | 14049 | 102 | 22 | 14173
  Idiopathic Short Stature (ISS) | 2844 | 27 | 5 | 2876
  All Other Diagnostic Groups Not Listed | 1226 | 96 | 5 | 1327
  Born Small for Gestational Age (SGA) | 1276 | 18 | 1 | 1295
  SHOX Deficiency (SHOX-D) | 576 | 126 | 3 | 705
  Turner Syndrome (TS) | 1870 | 42 | 1 | 1913
  Unknown | 383 | 46 | 40 | 469

OUTCOME MEASURES:

1. Primary Outcome: Type 2 Diabetes Mellitus in GH-treated Participants
Time Frame: Year 15
Population: All treated participants with available age and calculable follow-up time. The treated participants were not compared with untreated but with rates from general population registries. The untreated participants predominantly contained neoplasm or SHOX deficient diagnoses, therefore had significant baseline differences from treated participants.
Measure: Number; unit: Incident Cases
Arm/Group | Treated
Number analyzed (Participants) | 21448
Incident Cases
  Ages 0 to 9 | 1
  Ages 10 to 14 | 9
  Ages 15 to 19 | 8
Statistical Analysis 1: Comparison: Treated; Epidemiological comparison between incidence of type 2 diabetes in study versus general population registry data, stratified by age and ethnicity; Test type: Superiority or Other; Standardized Incidence Ratio = 3.77, 95% CI 2-sided [2.24 to 5.96]

2. Primary Outcome: Primary Malignancies in Participant Without Previous Cancer History
Description: Due to the small number of participants involved, untreated and unknown treatment groups, data was not provided and could not be calculated.
Time Frame: Year 15
Population: All treated participants with available age, gender, and at least one follow-up excluding participants with previous cancer cases. Due to the small number of participants involved, untreated and unknown treatment groups, data was not provided and could not be calculated.
Measure: Number; unit: Incident Cases
Groups:
- Treated: Participants treated with Humatrope for improvement of growth
  Humatrope (rDNA origin): Dose, frequency and duration at discretion of attending physician.
Arm/Group | Treated
Number analyzed (Participants) | 20146
Incident Cases | 14
Statistical Analysis 1: Comparison: Treated; Epidemiological comparison between incidence of primary malignancies in study versus general population registry data, stratified by age and gender; Test type: Superiority or Other; Standardized Incidence Ratio = 0.71, 95% CI 2-sided [0.39 to 1.20]

3. Primary Outcome: Final Height (FH) Gain by Diagnostic Group
Description: The standard deviation score (SDS) reports the number of standard deviations from the mean for age and sex for an individual measurement (normal range is -2 to +2 SDS). Height SDS is derived by subtracting the population mean from individual's height value and then dividing that difference by the population standard deviation. Greater height SDS values indicate greater height. Due to the small number of participants involved, untreated and unknown treatment groups, data was not provided and could not be calculated.
Time Frame: Baseline through Year 15
Population: All treated participants who reached final height (at least 1: closed epiphyses, height velocity <2 centimeters per year, or last bone age >14 years [girls] or >16 years [boys]) with baseline height SDS and final height available. Data was not provided for untreated and unknown treatment groups, and could not be calculated.
Measure: Mean (Standard Deviation); unit: standard deviation score
Groups:
- Treated: Participants treated with somatropin for improvement of growth
  Somatropin (rDNA origin): Dose, frequency and duration at discretion of attending physician.
Arm/Group | Treated
Number analyzed (Participants) | 5075
standard deviation score
  All Baseline Height | -2.42 (1.01)
  All Final Height | -1.18 (1.12)
  All Final Height Gain | 1.24 (1.08)
  GHD Baseline Height: number analyzed (Participants) | 3079
  GHD Baseline Height | -2.35 (1.04)
  GHD Final Height: number analyzed (Participants) | 3080
  GHD Final Height | -0.96 (1.12)
  GHD Final Height Gain: number analyzed (Participants) | 3079
  GHD Final Height Gain | 1.39 (1.14)
  TS Baseline Height: number analyzed (Participants) | 695
  TS Baseline Height | -2.65 (.089)
  TS Final Height: number analyzed (Participants) | 695
  TS Final Height | -1.70 (0.94)
  TS Final Height Gain: number analyzed (Participants) | 695
  TS Final Height Gain | 0.95 (0.82)
  ISS Baseline Height: number analyzed (Participants) | 552
  ISS Baseline Height | -2.37 (0.80)
  ISS Final Height: number analyzed (Participants) | 552
  ISS Final Height | -1.26 (0.96)
  ISS Final Height Gain: number analyzed (Participants) | 552
  ISS Final Height Gain | 1.10 (0.98)
  SHOX-D Baseline Height: number analyzed (Participants) | 131
  SHOX-D Baseline Height | -2.36 (0.79)
  SHOX-D Final Height: number analyzed (Participants) | 131
  SHOX-D Final Height | -1.50 (0.97)
  SHOX-D Final Height Gain: number analyzed (Participants) | 131
  SHOX-D Final Height Gain | 0.86 (0.91)
  SGA Baseline Height: number analyzed (Participants) | 265
  SGA Baseline Height | -2.57 (0.86)
  SGA Final Height: number analyzed (Participants) | 265
  SGA Final Height | -1.47 (0.84)
  SGA Final Height Gain: number analyzed (Participants) | 265
  SGA Final Height Gain | 1.11 (0.96)
  CRI Baseline Height: number analyzed (Participants) | 14
  CRI Baseline Height | -2.54 (0.90)
  CRI Final Height: number analyzed (Participants) | 14
  CRI Final Height | -1.66 (1.27)
  CRI Final Height Gain: number analyzed (Participants) | 14
  CRI Final Height Gain | 0.88 (0.81)
  Other Baseline Height: number analyzed (Participants) | 300
  Other Baseline Height | -2.70 (1.32)
  Other Final Height: number analyzed (Participants) | 300
  Other Final Height | -1.69 (1.33)
  Other Final Height Gain: number analyzed (Participants) | 300
  Other Final Height Gain | 1.01 (1.10)
  Unknown Baseline Height: number analyzed (Participants) | 39
  Unknown Baseline Height | -2.30 (1.02)
  Unknown Final Height: number analyzed (Participants) | 39
  Unknown Final Height | -1.54 (1.10)
  Unknown Final Height Gain: number analyzed (Participants) | 39
  Unknown Final Height Gain | 0.75 (0.83)

4. Secondary Outcome: Percentage of Participants With Defects in Genes Associated With Pituitary Development
Description: Percentage of participants with genetic defects associated with pituitary development. Genes included but were not limited to GH1, Growth hormone releasing hormone receptor (GHRHR), Homeobox gene expressed in embryonic stem cells (HESX1), LIM homeobox 3 (LHX3), POU domain, class 1, transcription factor 1 (POU1F1), and Prophet of Pit1 (PROP1).
Time Frame: Baseline through Year 15
Population: All SME participants (including treated, untreated, and unknown groups) with available results of DNA (deoxyribonucleic acid) analysis available and GHD diagnosis.
Measure: Number; unit: percentage of participants
Groups:
- Treated: Participants treated with somatropin for improvement of growth with a history of neoplasia or in those with any short stature homeobox (SHOX)-related disorder.
- Untreated: Participants not treated with a history of neoplasia or in those with any short stature homeobox (SHOX)-related disorder.
- Unknown: Treatment with somatropin unknown.
Arm/Group | Treated | Untreated | Unknown
Number analyzed (Participants) | 476 | 412 | 26
percentage of participants | 6.7 | 14.8 | 0.0

5. Secondary Outcome: Predicted First Year Height Gain Versus Actual First Year Height Gain
Description: The value for predicted and observed is of limited bearing, it is how each participant's predicted versus observed height gain compare and this is best estimated by the R-squared. An estimation parameter would not be a correct format for the R2 data. R2 can take value between 0 and 1 with values closer to 0 representing a poor fit while values closer to 1 representing a perfect fit
Time Frame: Baseline through Year 15
Population: All participants with predicted and actual first year height gain available and TS or GHD diagnosis. Data was not provided for untreated and unknown treatment groups, and could not be calculated.
Measure: Number; unit: R Squared
Arm/Group | Treated
Number analyzed (Participants) | 999
R Squared
  TS: number analyzed (Participants) | 115
  TS | 0.261
  GHD: number analyzed (Participants) | 884
  GHD | 0.408

6. Secondary Outcome: Change From Baseline to Final Height in Anthropometric Measures for Participants With SHOX Deficiency
Time Frame: Baseline, Year 15
Population: All SHOX-D Participants, GH-treated, with available height SDS at baseline and final height. Data was not provided for untreated and unknown treatment groups, and could not be calculated.
Measure: Mean (Standard Deviation); unit: standard deviation score
Arm/Group | Treated
Number analyzed (Participants) | 144
standard deviation score
  Height SDS | 0.8 (0.9)
  Sitting Height (SH) SDS: number analyzed (Participants) | 44
  Sitting Height (SH) SDS | 1.4 (1.0)
  Arm Span (AS) SDS: number analyzed (Participants) | 10
  Arm Span (AS) SDS | -0.6 (6.2)
  SH SDS/Height SDS: number analyzed (Participants) | 44
  SH SDS/Height SDS | -0.7 (1.8)
  AS SDS/Height SDS: number analyzed (Participants) | 10
  AS SDS/Height SDS | 1.0 (3.0)
  AS SDS/SH SDS: number analyzed (Participants) | 6
  AS SDS/SH SDS | 10.2 (22.9)

7. Secondary Outcome: Percentage of Participants With Recurrent Neoplasms and Second Neoplasms in Childhood Cancer Survivors
Description: Percentage of participants with recurrence/progression of primary neoplastic disease and/or development of secondary neoplasms in childhood cancer survivors.
Time Frame: Baseline through Year 15
Population: All SME, treated participants with previous neoplastic disease and at least one follow-up visit. Data was not provided for untreated and unknown treatment groups, and could not be calculated.
Measure: Number; unit: percentage of participants
Arm/Group | Treated
Number analyzed (Participants) | 1087
percentage of participants
  Recurrences | 6.81
  Second Neoplasms: number analyzed (Participants) | 622
  Second Neoplasms | 4.98

8. Secondary Outcome: Percentage of Participants With De Novo Neoplasms
Description: Percentage of participants with the development of de novo neoplastic disease with no history of prior neoplasia.
Time Frame: Baseline through Year 15
Population: All SME, GH-treated participants with at least one follow-up visit. Data was not provided for untreated and unknown treatment groups, and could not be calculated.
Measure: Number; unit: percentage of participants
Arm/Group | Treated
Number analyzed (Participants) | 20556
percentage of participants | 0.07

9. Secondary Outcome: Diabetes Mellitus (DM) in Somatropin-Treated Children With Different Short Stature Diagnoses
Time Frame: Baseline through Year 15
Population: All treated participants with available age and calculable follow-up time, and diabetes mellitus (DM), type 1 diabetes mellitus (T1) or type 2 diabetes mellitus (T2). Data was not provided for untreated and unknown treatment groups, and could not be calculated.
Measure: Number; unit: Incident Cases
Arm/Group | Treated
Number analyzed (Participants) | 21448
Incident Cases
  All DM | 38
  GHD DM: number analyzed (Participants) | 13507
  GHD DM | 22
  TS DM: number analyzed (Participants) | 1815
  TS DM | 6
  ISS DM: number analyzed (Participants) | 2645
  ISS DM | 4
  SHOX-D DM: number analyzed (Participants) | 564
  SHOX-D DM | 0
  SGA DM: number analyzed (Participants) | 1111
  SGA DM | 2
  Other DM: number analyzed (Participants) | 1488
  Other DM | 4
  Unknown DM: number analyzed (Participants) | 318
  Unknown DM | 0
  All T1 | 19
  GHD T1: number analyzed (Participants) | 13507
  GHD T1 | 10
  TS T1: number analyzed (Participants) | 1815
  TS T1 | 3
  ISS T1: number analyzed (Participants) | 2645
  ISS T1 | 3
  SHOX-D T1: number analyzed (Participants) | 564
  SHOX-D T1 | 0
  SGA T1: number analyzed (Participants) | 1111
  SGA T1 | 0
  Other T1: number analyzed (Participants) | 1488
  Other T1 | 3
  Unknown T1: number analyzed (Participants) | 318
  Unknown T1 | 0
  All T2 | 18
  GHD T2: number analyzed (Participants) | 13507
  GHD T2 | 12
  TS T2: number analyzed (Participants) | 1815
  TS T2 | 3
  ISS T2: number analyzed (Participants) | 2645
  ISS T2 | 0
  SHOX-D T2: number analyzed (Participants) | 564
  SHOX-D T2 | 0
  SGA T2: number analyzed (Participants) | 1111
  SGA T2 | 2
  Other T2: number analyzed (Participants) | 1488
  Other T2 | 1
  Unknown T2: number analyzed (Participants) | 318
  Unknown T2 | 0
Statistical Analysis 1: Comparison: Treated; Epidemiological comparison between incidence of type 2 diabetes in study versus general population registry data, stratified by age and ethnicity. Standardized Incidence Ratio for All DM (T1, T2 and DM Not Otherwise Specified [NOS] Combined); Test type: Superiority or Other; Standardized Incidence Ratio = 3.03, 95% CI 2-sided [2.14 to 4.15]
Statistical Analysis 2: Comparison: Treated; Epidemiological comparison between incidence of type 2 diabetes in study versus general population registry data, stratified by age and ethnicity. Standardized Incidence Ratio for GHD DM (T1, T2 and DM NOS Combined); Test type: Superiority or Other; Standardized Incidence Ratio = 2.74, 95% CI 2-sided [1.72 to 4.15]
Statistical Analysis 3: Comparison: Treated; Epidemiological comparison between incidence of type 2 diabetes in study versus general population registry data, stratified by age and ethnicity. Standardized Incidence Ratio for TS DM (T1, T2 and DM NOS Combined); Test type: Superiority or Other; Standardized Incidence Ratio = 4.91, 95% CI 2-sided [1.80 to 10.69]
Statistical Analysis 4: Comparison: Treated; Epidemiological comparison between incidence of type 2 diabetes in study versus general population registry data, stratified by age and ethnicity. Standardized Incidence Ratio for ISS DM (T1, T2 and DM NOS Combined); Test type: Superiority or Other; Standardized Incidence Ratio = 3.10, 95% CI 2-sided [0.84 to 7.93]
Statistical Analysis 5: Comparison: Treated; Epidemiological comparison between incidence of type 2 diabetes in study versus general population registry data, stratified by age and ethnicity. Standardized Incidence Ratio for SHOX-D DM (T1, T2 and DM NOS Combined); Test type: Superiority or Other; Standardized Incidence Ratio = 0.00, 95% CI 2-sided [0.00 to 11.83]
Statistical Analysis 6: Comparison: Treated; Epidemiological comparison between incidence of type 2 diabetes in study versus general population registry data, stratified by age and ethnicity. Standardized Incidence Ratio for SGA DM (T1, T2 and DM NOS Combined); Test type: Superiority or Other; Standardized Incidence Ratio = 3.00, 95% CI 2-sided [0.36 to 10.83]
Statistical Analysis 7: Comparison: Treated; Epidemiological comparison between incidence of type 2 diabetes in study versus general population registry data, stratified by age and ethnicity. Standardized Incidence Ratio for Other DM (T1, T2 and DM NOS Combined); Test type: Superiority or Other; Standardized Incidence Ratio = 4.55, 95% CI 2-sided [1.24 to 11.66]
Statistical Analysis 8: Comparison: Treated; Epidemiological comparison between incidence of type 2 diabetes in study versus general population registry data, stratified by age and ethnicity. Standardized Incidence Ratio for Unknown DM (T1, T2 and DM NOS Combined); Test type: Superiority or Other; Standardized Incidence Ratio = 0.00, 95% CI 2-sided [0.00 to 24.30]
Statistical Analysis 9: Comparison: Treated; Epidemiological comparison between incidence of type 2 diabetes in study versus general population registry data, stratified by age and ethnicity. Standardized Incidence Ratio for All T1 DM; Test type: Superiority or Other; Standardized Incidence Ratio = 0.92, 95% CI 2-sided [0.56 to 1.44]
Statistical Analysis 10: Comparison: Treated; Epidemiological comparison between incidence of type 2 diabetes in study versus general population registry data, stratified by age and ethnicity. Standardized Incidence Ratio for GHD T1DM; Test type: Superiority or Other; Standardized Incidence Ratio = 0.76, 95% CI 2-sided [0.36 to 1.40]
Statistical Analysis 11: Comparison: Treated; Epidemiological comparison between incidence of type 2 diabetes in study versus general population registry data, stratified by age and ethnicity. Standardized Incidence Ratio for TS T1DM; Test type: Superiority or Other; Standardized Incidence Ratio = 1.50, 95% CI 2-sided [0.31 to 4.38]
Statistical Analysis 12: Comparison: Treated; Epidemiological comparison between incidence of type 2 diabetes in study versus general population registry data, stratified by age and ethnicity. Standardized Incidence Ratio for ISS T1DM; Test type: Superiority or Other; Standardized Incidence Ratio = 1.42, 95% CI 2-sided [0.29 to 4.14]
Statistical Analysis 13: Comparison: Treated; Epidemiological comparison between incidence of type 2 diabetes in study versus general population registry data, stratified by age and ethnicity. Standardized Incidence Ratio for SHOX-D T1DM; Test type: Superiority or Other; Standardized Incidence Ratio = 0.00, 95% CI 2-sided [0.00 to 7.23]
Statistical Analysis 14: Comparison: Treated; Epidemiological comparison between incidence of type 2 diabetes in study versus general population registry data, stratified by age and ethnicity. Standardized Incidence Ratio for SGA T1DM; Test type: Superiority or Other; Standardized Incidence Ratio = 0.00, 95% CI 2-sided [0.00 to 3.38]
Statistical Analysis 15: Comparison: Treated; Epidemiological comparison between incidence of type 2 diabetes in study versus general population registry data, stratified by age and ethnicity. Standardized Incidence Ratio for Other T1DM; Test type: Superiority or Other; Standardized Incidence Ratio] = 2.09, 95% CI 2-sided [0.43 to 6.10]
Statistical Analysis 16: Comparison: Treated; Epidemiological comparison between incidence of type 2 diabetes in study versus general population registry data, stratified by age and ethnicity. Standardized Incidence Ratio for Unknown T1DM; Test type: Superiority or Other; Standardized Incidence Ratio] = 0.00, 95% CI 2-sided [0.00 to 14.84]
Statistical Analysis 17: Comparison: Treated; Epidemiological comparison between incidence of type 2 diabetes in study versus general population registry data, stratified by age and ethnicity. Standardized Incidence Ratio for All T2 DM; Test type: Superiority or Other; Standardized Incidence Ratio = 3.79, 95% CI 2-sided [2.24 to 5.96]
Statistical Analysis 18: Comparison: Treated; Epidemiological comparison between incidence of type 2 diabetes in study versus general population registry data, stratified by age and ethnicity. Standardized Incidence Ratio for GHD T2DM; Test type: Superiority or Other; Standardized Incidence Ratio = 3.93, 95% CI 2-sided [2.03 to 6.87]
Statistical Analysis 19: Comparison: Treated; Epidemiological comparison between incidence of type 2 diabetes in study versus general population registry data, stratified by age and ethnicity. Standardized Incidence Ratio for TS T2DM; Test type: Superiority or Other; Standardized Incidence Ratio = 6.46, 95% CI 2-sided [1.33 to 18.89]
Statistical Analysis 20: Comparison: Treated; Epidemiological comparison between incidence of type 2 diabetes in study versus general population registry data, stratified by age and ethnicity. Standardized Incidence Ratio for ISS T2DM; Test type: Superiority or Other; Standardized Incidence Ratio = 0.00, 95% CI 2-sided [0.00 to 7.52]
Statistical Analysis 21: Comparison: Treated; Epidemiological comparison between incidence of type 2 diabetes in study versus general population registry data, stratified by age and ethnicity. Standardized Incidence Ratio for SHOX-D T2DM; Test type: Superiority or Other; Standardized Incidence Ratio = 0.00, 95% CI 2-sided [0.00 to 31.16]
Statistical Analysis 22: Comparison: Treated; Epidemiological comparison between incidence of type 2 diabetes in study versus general population registry data, stratified by age and ethnicity. Standardized Incidence Ratio for SGA T2DM; Test type: Superiority or Other; Standardized Incidence Ratio = 7.90, 95% CI 2-sided [0.96 to 28.52]
Statistical Analysis 23: Comparison: Treated; Epidemiological comparison between incidence of type 2 diabetes in study versus general population registry data, stratified by age and ethnicity. Standardized Incidence Ratio for Other T2DM; Test type: Superiority or Other; Standardized Incidence Ratio = 3.00, 95% CI 2-sided [0.08 to 16.70]
Statistical Analysis 24: Comparison: Treated; Epidemiological comparison between incidence of type 2 diabetes in study versus general population registry data, stratified by age and ethnicity. Standardized Incidence Ratio for Unknown T2DM; Test type: Superiority or Other; Standardized Incidence Ratio = 0.00, 95% CI 2-sided [0.00 to 63.97]

ADVERSE EVENTS:
Groups:
- Untreated: No treatment with somatropin in participants with a history of neoplasia or in those with any SHOX deficiency-related disorder.
- EG002: Treatment with Humatrope unknown.
Arm/Group | Treated | Untreated | EG002
Serious Adverse Events (participants affected / at risk) | 547/21177 | 14/306 | 0/40
Other Adverse Events (participants affected / at risk) | 6180/21177 | 126/306 | 0/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Treated (N=21177) | Untreated (N=306) | EG002 (N=40)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 0 (0) | 0 (0)
Aplastic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (2) | 0 (0)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac disorder (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary valve disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Arnold-chiari malformation (Congenital, familial and genetic disorders) | 2 (2) | 0 (0) | 0 (0)
Brachydactyly (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Coarctation of the aorta (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Congenital aplastic anaemia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Cryptorchism (Congenital, familial and genetic disorders) | 2/12692 (2) | 0 (0) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 1/12692 (1) | 0 (0) | 0 (0)
Imperforate hymen (Congenital, familial and genetic disorders) | 1/8458 (1) | 0 (0) | 0 (0)
Intestinal malrotation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Laryngomalacia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Oculoauriculovertebral dysplasia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Prader-willi syndrome (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Rathke's cleft cyst (Congenital, familial and genetic disorders) | 1 (2) | 0 (0) | 0 (0)
Tourette's disorder (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular septal defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Middle ear disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Tympanic membrane disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 5 (6) | 0 (0) | 0 (0)
Adrenocortical insufficiency acute (Endocrine disorders) | 10 (13) | 0 (0) | 0 (0)
Diabetes insipidus (Endocrine disorders) | 4 (4) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Precocious puberty (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Secondary adrenocortical insufficiency (Endocrine disorders) | 3 (3) | 0 (0) | 0 (0)
Secondary hypogonadism (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Deformity of orbit (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Iridocyclitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Keratoconus (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Oculogyric crisis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Papilloedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 3 (3) | 0 (0) | 0 (0)
Strabismus (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Uveitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 5 (5) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0)
Oesophageal rupture (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Volvulus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 16 (22) | 0 (0) | 0 (0)
Asthenia (General disorders) | 2 (2) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cyst (General disorders) | 2 (2) | 0 (0) | 0 (0)
Death (General disorders) | 4 (4) | 0 (0) | 0 (0)
Device malfunction (General disorders) | 2 (3) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 2 (2) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 6 (8) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 2 (2) | 0 (0) | 0 (0)
Anaphylactoid reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Kidney transplant rejection (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 14 (14) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Brain abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Catheter site cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Cellulitis orbital (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cholangitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 17 (18) | 0 (0) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
H1n1 influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Haemophilus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hepatitis a (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hepatitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster disseminated (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 7 (7) | 0 (0) | 0 (0)
Latent tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lymph node tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Mastoiditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Meningitis aseptic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Meningitis bacterial (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Meningitis viral (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Mycoplasma infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Otitis media chronic (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Parotitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 22 (28) | 1 (1) | 0 (0)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 7 (7) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 2 (11) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rotavirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 5 (5) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Shunt infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 5 (5) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 7 (7) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Varicella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 9 (11) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 6 (6) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 0 (0)
Hepatic rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 6 (6) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Radiation injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 6 (6) | 0 (0) | 0 (0)
Shunt malfunction (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Shunt occlusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Splenic injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Splenic rupture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Sports injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Traumatic renal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Body temperature fluctuation (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Insulin-like growth factor increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Salmonella test positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 8 (10) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 18 (23) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Polydipsia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Tetany (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 6 (6) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Weight gain poor (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bone cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bone development abnormal (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bone disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bone lesion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Epiphysiolysis (Musculoskeletal and connective tissue disorders) | 11 (12) | 0 (0) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Extremity contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Kyphoscoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Kyphosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Limb asymmetry (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Limb deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Posture abnormal (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 10 (10) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0)
Anaplastic astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1) | 0 (0)
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Choroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Craniopharyngioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 19 (22) | 0 (0) | 0 (0)
Ependymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Ewing's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Fibrous cortical defect (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Inflammatory pseudotumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Medulloblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0) | 0 (0)
Medulloblastoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Neoplasm recurrence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 0 (0)
Neuroblastoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Neurofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Optic glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Osteochondroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Osteoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Osteosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/8458 (1) | 0 (0) | 0 (0)
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/8458 (1) | 0 (0) | 0 (0)
Pancreatic neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Peripheral nerve sheath tumour malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pituitary tumour recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Primitive neuroectodermal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prolactinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Testicular germ cell cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/12692 (1) | 0 (0) | 0 (0)
Tongue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Acquired epileptic aphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Benign intracranial hypertension (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Conus medullaris syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dyslalia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0)
Facial paresis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 8 (8) | 1 (2) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hemiplegic migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemic seizure (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Infantile spasms (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Intraventricular haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Meningism (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Migraine with aura (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Moyamoya disease (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0)
Myoclonus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraplegia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Partial seizures (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Peroneal nerve palsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Petit mal epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 16 (17) | 2 (2) | 0 (0)
Status epilepticus (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tethered cord syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Unresponsive to stimuli (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Visual field defect (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Anger (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Anorexia nervosa (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0)
Asperger's disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Conversion disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Eating disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Mental disorder (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Obsessive-compulsive disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Phobia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Reactive attachment disorder of infancy or early childhood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicidal behaviour (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Anuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 5 (5) | 0 (0) | 0 (0)
Glomerulonephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Post streptococcal glomerulonephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Fallopian tube cyst (Reproductive system and breast disorders) | 1/8458 (1) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 1/8458 (1) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 2/8458 (2) | 0 (0) | 0 (0)
Testicular torsion (Reproductive system and breast disorders) | 2/12692 (2) | 0 (0) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 0 (0) | 0 (0)
Allergic respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 0 (0) | 0 (0)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pulmonary artery dilatation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0) | 0 (0)
Snoring (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tonsillar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Purpura fulminans (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Puberty (Social circumstances) | 1 (1) | 0 (0) | 0 (0)
Adenoidectomy (Surgical and medical procedures) | 3 (3) | 0 (0) | 0 (0)
Adenotonsillectomy (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0)
Arthrodesis (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Bone marrow transplant (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Cleft lip repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Ear operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Eye operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Hydrocele operation (Surgical and medical procedures) | 1/12692 (1) | 0 (0) | 0 (0)
Inguinal hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Jejunostomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Leg amputation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Limb operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Medical device implantation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Meningioma surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Nasal septal operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Oesophagogastric fundoplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Oophorectomy bilateral (Surgical and medical procedures) | 1/8458 (1) | 0 (0) | 0 (0)
Orchidectomy (Surgical and medical procedures) | 1/12692 (1) | 0 (0) | 0 (0)
Orchidopexy (Surgical and medical procedures) | 2/12692 (2) | 0 (0) | 0 (0)
Osteotomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Renal transplant (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0)
Salpingo-oophorectomy bilateral (Surgical and medical procedures) | 1/8458 (1) | 0 (0) | 0 (0)
Scoliosis surgery (Surgical and medical procedures) | 2 (3) | 0 (0) | 0 (0)
Spinal fusion surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Tenotomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Tonsillectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Ventriculo-peritoneal shunt (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0)
Wisdom teeth removal (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Angiodysplasia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.2% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Treated (N=21177) | Untreated (N=306) | EG002 (N=40)
Turner's syndrome (Congenital, familial and genetic disorders) | 19/8458 (19) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 99 (100) | 3 (3) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 48 (50) | 2 (2) | 0 (0)
Delayed puberty (Endocrine disorders) | 192 (193) | 3 (3) | 0 (0)
Diabetes insipidus (Endocrine disorders) | 49 (49) | 1 (1) | 0 (0)
Hypogonadism (Endocrine disorders) | 129 (131) | 0 (0) | 0 (0)
Hypopituitarism (Endocrine disorders) | 85 (85) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 391 (391) | 2 (2) | 0 (0)
Precocious puberty (Endocrine disorders) | 262 (266) | 11 (11) | 0 (0)
Primary hypothyroidism (Endocrine disorders) | 193 (195) | 7 (7) | 0 (0)
Secondary hypogonadism (Endocrine disorders) | 97 (97) | 4 (4) | 0 (0)
Secondary hypothyroidism (Endocrine disorders) | 312 (314) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 133 (147) | 11 (16) | 0 (0)
Constipation (Gastrointestinal disorders) | 147 (153) | 13 (17) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 69 (74) | 13 (14) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 57 (58) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 65 (71) | 12 (17) | 0 (0)
Vomiting (Gastrointestinal disorders) | 115 (138) | 5 (6) | 0 (0)
Asthenia (General disorders) | 53 (55) | 0 (0) | 0 (0)
Fatigue (General disorders) | 73 (77) | 14 (16) | 0 (0)
Injection site pain (General disorders) | 53 (55) | 0 (0) | 0 (0)
No adverse event (General disorders) | 110 (110) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 118 (148) | 5 (12) | 0 (0)
Hypersensitivity (Immune system disorders) | 44 (45) | 0 (0) | 0 (0)
Multiple allergies (Immune system disorders) | 70 (70) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 99 (104) | 7 (7) | 0 (0)
Bronchitis (Infections and infestations) | 90 (112) | 2 (3) | 0 (0)
Ear infection (Infections and infestations) | 70 (89) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 123 (140) | 5 (5) | 0 (0)
Influenza (Infections and infestations) | 108 (131) | 4 (5) | 0 (0)
Nasopharyngitis (Infections and infestations) | 78 (108) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 199 (264) | 10 (15) | 0 (0)
Pharyngitis (Infections and infestations) | 51 (55) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 70 (82) | 4 (5) | 0 (0)
Pneumonia (Infections and infestations) | 62 (74) | 3 (4) | 0 (0)
Sinusitis (Infections and infestations) | 99 (111) | 8 (10) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 199 (279) | 20 (33) | 0 (0)
Urinary tract infection (Infections and infestations) | 49 (58) | 4 (5) | 0 (0)
Varicella (Infections and infestations) | 43 (44) | 1 (1) | 0 (0)
Blood corticotrophin decreased (Investigations) | 51 (51) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 64 (66) | 5 (5) | 0 (0)
Vitamin d deficiency (Metabolism and nutrition disorders) | 135 (143) | 36 (40) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 373 (425) | 16 (23) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 87 (92) | 7 (7) | 0 (0)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 52 (52) | 1 (1) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 58 (59) | 7 (7) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 111 (128) | 10 (17) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 412 (416) | 8 (8) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 129 (134) | 5 (5) | 0 (0)
Dizziness (Nervous system disorders) | 43 (45) | 6 (11) | 0 (0)
Headache (Nervous system disorders) | 594 (680) | 36 (67) | 0 (0)
Migraine (Nervous system disorders) | 63 (64) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 87 (89) | 4 (4) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 43 (43) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 65 (65) | 10 (10) | 0 (0)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 389 (389) | 5 (5) | 0 (0)
Depression (Psychiatric disorders) | 81 (81) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 47 (48) | 4 (4) | 0 (0)
Enuresis (Renal and urinary disorders) | 95 (101) | 2 (2) | 0 (0)
Amenorrhoea (Reproductive system and breast disorders) | 21/8458 (21) | 1/166 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 16/8458 (16) | 4/166 (6) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 87/12692 (89) | 0 (0) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 23/8458 (23) | 2/166 (2) | 0 (0)
Ovarian failure (Reproductive system and breast disorders) | 85/8458 (85) | 7/166 (7) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 174 (180) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 70 (75) | 5 (6) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 38 (40) | 6 (9) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 61 (69) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 55 (55) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 130 (135) | 5 (5) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 73 (75) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 47 (48) | 7 (9) | 0 (0)
Hypertension (Vascular disorders) | 45 (47) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days